CLINICAL TRIAL: NCT05782894
Title: A Multicenter, Randomized, Single-blinded, Parallel, Two-step Trial to Evaluate the Effectiveness and Safety of Remimazolam Besylate for Injection for Sedation in ICU Patients
Brief Title: Step 2 of A Two-step Trial to Evaluate the Effectiveness and Safety of Remimazolam Besylate for Sedation in ICU Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Yichang Humanwell Pharmaceutical Co., Ltd., China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WHUICU202208
Record Dates: First submitted 2023-02-18; First posted 2023-03-24 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-12

CONDITIONS: Sedative; Mechanical Ventilation
MeSH Terms: interventions — Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam besylate (Experimental): Remimazolam besylate
  Interventions: Drug: Remimazolam besylate; Drug: Remifentanil
- Propofol (Active Comparator): Propofol
  Interventions: Drug: Propofol; Drug: Remifentanil

INTERVENTIONS:
Drug: Remimazolam besylate — 0~2.0mg/kg/h
  Arms: Remimazolam besylate
Drug: Propofol — 0.3~4.0mg/kg/h
  Arms: Propofol
Drug: Remifentanil — 1.5~12μg/kg/h

SUMMARY:
A randomized non-inferior trial comparing remimazolam besylate with propofol for short-term sedation during invasive mechanical ventilation in intensive care units

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years
* Body mass index (BMI) ≥18 and ≤ 30 kg/m2
* Being Intubated and mechanically ventilated ≤48 hours before enrollment and expected to be on ventilator for at least 6 hours
* Requirement for light to moderate sedation (a Richmond agitation-sedation scale score of -2 to 1)

Exclusion Criteria:

* Refusal to be included
* Allergy or unsuitability to any composition of study drugs or remifentanil
* Living expectancy less than 48 hours
* Myasthenia gravis
* Status asthmaticus
* Abdominal compartment syndrome
* Serious hepatic dysfunction (CTP 10-15);
* Chronic kidney disease with glomerular filtration rate (GFR) < 29 ml/min/1.73m2
* Mean blood pressure less than 65 mm Hg or the need of a continuous infusion of norepinephrine at ≥0.5 ug/kg/min to maintain Mean blood pressure ≥ 65 mm Hg
* Possible requirement for surgery or bedside tracheostomy in 24 hours
* Possible requirement for renal replacement therapy in 24 hours
* Acute severe neurological disorder and any other condition interfering with sedation assessment
* Abuse of controlled substances or alcohol
* Pregnancy or lactation
* Inclusion in another interventional trial in the past 30 days
* Other conditions deemed unsuitable to be included

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Successful sedation | 24 hours
  70% of time in the target sedation range in participants without rescue sedation

SECONDARY OUTCOMES:
The percentage of time in the target sedation range without rescue sedation | 24 hours
  The percentage of time in the target sedation range without rescue sedation
Number of patients needing rescue sedation | 24 hours
  Whether participants need sedative drugs other than the study drug to re maintain targeted sedation level
Number of patients needing repeated boluses of the study drug | 24 hours
  Whether participants need repeated boluses of the study durg other than the loading dose to maintain targeted sedation level
The amount of remifentanil in ug/kg/h | 24 hours
  The amount of remifentanil in ug/kg/h used in each patient in both groups

OTHER OUTCOMES:
Hypotension | 24 hours
  Whether hypotension occurs in participants
Delirium | 24 hours
  Whether delirium occurs in participants

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Tang Y, Shu H, Ren L, Li R, Zou X, Qi H, Ouyang Y, Wu Y, Xu J, Fang X, Yang X, Shang Y. Remimazolam Besylate Versus Propofol for Short-Term Sedation in Critically Ill Patients Receiving Mechanical Ventilation: Protocol for a Multicenter Randomized Non-inferior Trial. Adv Ther. 2025 Aug;42(8):4081-4088. doi: 10.1007/s12325-025-03268-7. Epub 2025 Jun 10. PMID 40493335